CLINICAL TRIAL: NCT03199495
Title: Efficacy of Electroacupuncture on Acute Abdomen Emergency Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Lee Tsung Chieh, Vice director of Chinese Medicine, Changhua Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChanghuaCH
Record Dates: First submitted 2017-06-13; First posted 2017-06-27 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Acupuncture
Keywords: traditional Chinese medicine; electroacupuncture; abdominal pain
MeSH Terms: conditions — Abdominal Pain | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupuncture (Experimental): Participants were randomized divided into experimental and control groups .Acupuncture included Hegu (LI 4), Neiguan (PC6), Zusali (ST 36), Shanjuxu (ST37), Xiajuxu (ST39), Taichong (LR3) and Taibai(SP3) on both hands and legs. Acupuncture included Hegu (LI 4) and Neiguan (PC6), Zusali (ST 36) and Taichong (LR3) with electrical stimulation were conducted. The frequency of electrical stimulation was 2 Hz and the intensities of the stimulation was below 9.8 mA for 15 minutes.After 15 minutes treatment, acupuncture were removed and after 15 minutes the investigators stated to evaluate.
  Interventions: Other: electroacupuncture
- sham electroacupuncture (Sham Comparator): Participants were randomized divided into experimental and control groups. The Vaccaria Seeds (scientific name:Vaccaria segetalis) will be applied in control group. Vaccaria Seed is a spherical, smooth and hard seed, which is commonly used on ear acupuncture point. In control group, Vaccaria Seeds will be secured on the acupuncture point the same as experimental group, and coverd by transcutaneous electrical nerve stimulation (TENS), which is actually not turned on. The intervention will last for 15 minutes.After 15 minutes treatment, acupuncture were removed and after 15 minutes the investigators stated to evaluate.
  Interventions: Other: electroacupuncture

INTERVENTIONS:
Other: electroacupuncture — acupuncture needle with TENS device

SUMMARY:
Contrast to conventional Western medicine, traditional Chinese medicine is the most common used therapy of complementary and alternative medicine. Taiwan inherits traditional Chinese culture, and the people popularly accept traditional Chinese medicine for general diseases. However, most patients with acute or critical illness are used to admit to emergency department for medical services, and then transfer to the department of related specialist for further treatment. During the course of staying at emergent observation room, some diseases do not meet the criteria of admission and keep for evaluation. The longer of staying at emergent observation room the more waste medical resources.

The Chinese medicine department of Changhua Christian hospital has treated patients, who consulted us at their own dispense, with subjective discomfort but remained at the emergent observation room. Detailed contents of this study include the Chinese and Western medicine, pharmaceutical, nursing cooperation mode, monitoring clinical effect of treating of the patients diagnosed with intestinal obstruction or ileus who complain about nausea, vomiting, abdominal pain, abdominal distension or constipation.And the patients were assigned to the control and treatment group. Then we give the treatment group with the electroacupuncture treatment,and the control groupe with the Chinese medicine seeds and the transcutaneous nerve stimulation (no power).The patients were diagnosed with objective analysis of tongue diagnosis, pulse diagnosis, heart rate variability, and questionnaire of pain. Hope that we can assess the efficacy of both two different treatment,and also assess the cost of medical care, and try to complete the syndromes statistical analysis of traditional Chinese medicine for abdominal pain, building the relevance of Chinese medicine physical assessment teaching and clinical efficacy.

The most important of this clinical teaching is that, this is a good opportunity for Chinese medicine and Western medicine to cooperate with each other at the emergency department to confirm the efficacy of traditional Chinese medicine, not only in the field of chronic or geriatric diseases, but also in the field of emergency with the evidence base. This factually achieves communication and integration of Chinese and Western medicine, and benefits the public.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 20-90 years old,who accepted to enter this trial
2. The patients diagnosed with intestinal obstruction or ileus who complain about nausea, vomiting, abdominal pain, abdominal distension or constipation.
3. ICD-10 is R101-R1012

Exclusion Criteria:

Does not meet the above conditions

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Assessed the change of pain | Before intervention/ 15 minutes after intervention/ 3 days after the intervention
  The primary outcome evaluation was the visual analog scale (VAS) for pain. Visual analog scale is graded from 0 (no pain) to 10 (worst possible pain) and has proven its usefulness and clinical validity for the evaluation of pain. Patients were evaluated at two timepoints in this study: intervention (VAS-1), after intervention (VAS-2), 3 days after the intervention (VAS-3).
Assessed the change of pain | Before intervention/ 15 minutes after intervention/ 3 days after the intervention
  The primary outcome evaluation was the the brief pain inventory (BPI) for pain. Brief pain inventory is used to assess the severity of pain and the impact of pain on daily functions. Patients were evaluated at two timepoints in this study: intervention (BPI-1), after intervention (BPI-2), 3 days after the intervention (BPI-3).

SECONDARY OUTCOMES:
The duration that patient stay at emergency department (ED) . | The duration is from the post-treatment to after 3 days that the participant may be discharged.
  The investigators will keep track of the direction (conditions) of post-treatment participant, their time duration at Emergency Department Observation sections.
The ratio is that patient goes to emergency department (ED) because of the same chief complain unexpectedly. | The duration is from the post-treatment to after 3 days that the participant may be discharged.
  The investigators will keep track of the rate of post-treatment participant of return to the emergency department (ED) for the same chief complain within 3 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital, Changhua, Changhua County, Taiwan

REFERENCES:
- [Derived] Chang YY, Chiu CW, Chen CY, Chang CF, Lee TC, Lo LC, Lee CY, Chang K, Chen PW, Hsieh CJ, Chang YJ, Huang SY. Efficacy of electroacupuncture on acute abdomen emergency care: study protocol for a randomized controlled trial. Trials. 2020 Feb 24;21(1):224. doi: 10.1186/s13063-020-4071-3. PMID 32093785